CLINICAL TRIAL: NCT00615238
Title: Physical Activity in the Treatment of Obesity: A Randomized Trial
Brief Title: Physical Activity in the Treatment of Obesity
Acronym: CHANGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DK53907 (completed 2004); R01DK053907 (NIH)
Record Dates: First submitted 2008-02-12; First posted 2008-02-14 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2010-03

CONDITIONS: Obesity
Keywords: overweight, physical activity, body composition, metabolic syndrome
MeSH Terms: conditions — Obesity; Overweight; Motor Activity; Metabolic Syndrome | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diet plus continuous bouts (Experimental): diet-plus-continuous bouts of vigorous aerobic exercise
  Interventions: Behavioral: Diet plus continuous bouts
- Diet plus short bouts (Experimental): diet-plus-short bouts of vigorous aerobic exercise accumulated throughout the day
  Interventions: Behavioral: Diet plus short bouts
- Diet plus moderate lifestyle activity (Experimental): diet-plus-moderate intensity lifestyle activity accumulated throughout the day
  Interventions: Behavioral: Diet plus moderate lifestyle activity

INTERVENTIONS:
Behavioral: Diet plus continuous bouts — Patients consumed a 1200 kcal/d diet and were instructed to perform 4 30-60 minute aerobic workouts per week
  Arms: Diet plus continuous bouts
Behavioral: Diet plus short bouts — Patients consumed a 1200 kcal/d diet and were instructed to perform short 10 minutes bouts of aerobic exercise 4 times per week
  Arms: Diet plus short bouts
Behavioral: Diet plus moderate lifestyle activity — Patients consumed a 1200 kcal/d diet and were instructed to accumulate moderate intensity physical activity on most days of the week.
  Arms: Diet plus moderate lifestyle activity

SUMMARY:
Although exercise is widely regarded as a key component in obesity treatment, few individuals seem able to adhere to exercise programs over time. In response, efforts have focused on developing new approaches to physical activity that may appeal to sedentary overweight persons. For instance, is has been shown that accumulating multiple short bouts of vigorous exercise may enhance both exercise adherence and weight loss in overweight persons. Accumulating moderate-intensity activity throughout the day may offer comparable health and weight benefits as a traditional exercise program. Public health recommendations now include the option of accumulating 30 minutes of moderate-intensity lifestyle activity for health and well-being. While these two options offer a viable alternative to those who dislike or cannot sustain continuous vigorous exercise programs, it is unclear whether the flexibility of accumulating physical activity or the vigorous intensity of the exercise is responsible for improved weight loss and long-term adherence.

The goal of this research is to extend our preliminary findings suggesting that moderate intensity lifestyle activity is an important and viable alternative to traditional structured vigorous exercise for obese dieting individuals. The primary specific aim of this project is to compare the effects of three modes of exercise on long-term weight regain. Participants will be 165 overweight men and women who are sedentary, but otherwise healthy. All participants will receive the same 16-week behavioral weight loss program and will be randomized to one of three exercise study conditions: 1) diet-plus-continuous bouts of vigorous aerobic exercise; 2) diet-plus-short bouts of vigorous aerobic exercise accumulated throughout the day; or 3) diet-plus-moderate intensity lifestyle activity accumulated throughout the day. By varying both the intensity and duration of exercise bouts, we can determine which type of exercise is associated with optimal outcomes one year later. Additional questions of interest include:

1. Does mode of exercise influence exercise adherence?
2. Does mode of exercise improve cardiovascular risk profiles similarly in all three conditions?
3. Does mode of exercise influence changes in body composition?
4. Does mode of exercise influence exercise enjoyment and exercise self-efficacy?

ELIGIBILITY:
Inclusion Criteria:Sedentary and >30 pounds above healthy weight. No plans to move from area for next 1.5 years. No plans for excessive travel.

-

Exclusion Criteria: recent weight loss or regular exercise (≥2 bouts per week), serious medical or psychiatric condition (cardiovascular, metabolic or orthopedic) or history of clinical depression or eating disorder.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2000-04; Primary Completion 2004-03 (Actual); Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
Participants were randomized to one of three diet and exercise study conditions. We were interested in which type of exercise is associated with optimal short- and long-term body composition changes. | Baseline, Week-16, Week-68

SECONDARY OUTCOMES:
Does mode of exercise improve cardiovascular risk profiles similarly in all three conditions? | Baseline, week-16, week-68

CONTACTS AND LOCATIONS:
Overall Officials: Jeremey D Walston, MD, Study Director — JHU School of Med; Susan J Bartlett, PhD, Study Director — JHU School of Med
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States